CLINICAL TRIAL: NCT03693950
Title: A Double-blind, Randomized, Controlled Clinical Study of the Pharmacokinetics, Pharmacodynamics, Tolerability, and Safety of Multiple Intravenous Injections of BCD-066 and Aranesp® in Healthy Volunteers
Brief Title: The Study of PK, PD, Safety of Multiple Intravenous Injections of BCD-066 and Aranesp in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BCD-066-3
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Results first posted 2019-07-01 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-066 1 µg/kg (Experimental): Healthy volunteers will receive BCD-066 1 μg/kg as weekly IV injections on Day 1, Day 8, Day 15, and Day 22.
  Interventions: Biological: BCD-066
- Aranesp 1 µg/kg (Active Comparator): Healthy volunteers will receive Aranesp 1 μg/kg as weekly IV injections on Day 1, Day 8, Day 15, and Day 22.
  Interventions: Biological: Aranesp

INTERVENTIONS:
Biological: BCD-066 — BCD-066 will be administered once a week intravenously in a dose 1 µg/kg
  Other Names: darbepoetin alfa
  Arms: BCD-066 1 µg/kg
Biological: Aranesp — Aranesp will be administered once a week intravenously in a dose 1 µg/kg
  Other Names: darbepoetin alfa
  Arms: Aranesp 1 µg/kg

SUMMARY:
BCD-066 is a darbepoetin alfa. Clinical study BCD-066-3 is a double-blind controlled, randomized, parallel-group study of the pharmacokinetics, pharmacodynamics, tolerability, and safety of multiple intravenous injections of BCD-066 and Aranesp®.

The purpose of the study is to confirm the equivalent pharmacokinetics, pharmacodynamics, safety, and tolerability of multiple IV injections of BCD-066 and Aranesp® in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Men from 18 to 45 years old (inclusive)
3. BMI within the normal limits (18.5 to 30 kg/m2)
4. Hemoglobin from 120 g/L to 150 g/L and hematocrit 41% to 49% at screening (before the first injection)
5. Serum transferring 2.15 g/L to 3.6 g/L; serum ferritin from 20 μg/L to 250 μg/L
6. Vitamin B12 from 187 pcg/mL to 883 pcg/mL; folic acid from 3.1 ng/mL to 20.5 ng/mL
7. Endogenous serum erythropoietin < 30 mIU/mL at screening
8. The subject is verified as "Healthy" according to results of standard clinical, laboratory and instrumental tests
9. Subject's ability (in the investigator's opinion) to follow the protocol procedures
10. The subject and his sexual partner with retained childbearing potential consent to implement reliable contraceptive methods starting 2 weeks before inclusion in the study and up to 2 weeks after the last dose of the test/reference drug. This requirement does not apply to surgically sterile subjects. Reliable contraception methods mean one barrier method in combination with one of the following: spermicides, intrauterine device and/or oral contraceptives used by the subject's partner.
11. The subject agrees not to drink alcohol for 24 h prior to each injection of the test/reference drug and for 72 h after the injection.

Exclusion Criteria:

1. Psychiatric disorders or other conditions that can affect the ability of the subject to follow the study protocol 2. Acute infections within 4 weeks before the study start 3. Results of laboratory and/or instrumental tests are outside the normal range 4. Chronic cardiovascular, bronchial and/or pulmonary, neuroendocrine GI, liver, kidney, and blood diseases, including ischemic heart disease, arterial hypertension, peripheral vascular and/or cerebral vascular disorders, and thrombocytosis 5. A history of chronic hemorrhages

-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD
Locations (1):
- BIOCAD, Saint Petersburg, Strelna, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Started | 29 | 28
Completed | 28 | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [22 to 31] | 27.50 [24 to 31] | 27.50 [24 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 28 | 28 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-72)
Description: The area concentration curve for darbepoetin alfa from injection to 72 h (AUC(0-72) after the first and the fourth IV injection of BCD-066 or Aranesp
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose
Measure: Median (Inter-Quartile Range); unit: pg/ml·h
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
pg/ml·h | 328215.65 [275530.49 to 401053.38] | 290827.12 [252607.47 to 349760.35]

2. Secondary Outcome: Cmax
Description: The maximum concentration of darbepoetin alfa in the serum after the first and the fourth IV injection of BCD-066 or Aranesp®
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose post-dose
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
pg/ml | 18365.15 [16861.5 to 22490] | 17003.25 [13716.6 to 19664.2]

3. Secondary Outcome: T½
Description: The elimination half-life
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
hours | 12.53 [11.334 to 13.235] | 12.69 [11.47 to 13.555]

4. Secondary Outcome: AUC(0-∞)
Description: The total area under the concentration curve from 0 to infinity
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose
Measure: Median (Inter-Quartile Range); unit: pg/ml·h
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
pg/ml·h | 331725.75 [276986.83 to 404075.52] | 296135.38 [260610.81 to 356012.29]

5. Secondary Outcome: Tmax
Description: The time to maximum drug concentration in the serum
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
hours | 0.125 [0.083 to 0.25] | 0.083 [0.083 to 0.25]

6. Secondary Outcome: Kel
Description: The elimination constant: kel=1/MRT, where MRT is median residence time: MRT=AUMC(0-72)/AUC(0-72)
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose
Measure: Median (Inter-Quartile Range); unit: fraction of drug per hour
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
fraction of drug per hour | 0.055 [0.052 to 0.06] | 0.055 [0.051 to 0.06]

7. Secondary Outcome: CL
Description: The total clearance
Time Frame: 5 min, 10 min, 15 min, 20 min, 30 min, 45 min, 1 h, 2 h, 4 h, 8 h, 16 h, 24 h, 48 h, 72 h post-dose
Measure: Median (Inter-Quartile Range); unit: ml/h
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
Number analyzed (Participants) | 28 | 28
ml/h | 230.358 [210.737 to 275.827] | 243.055 [197.849 to 299.107]

ADVERSE EVENTS:
Time Frame: AEs where collected from the first drug administration (visit 1, day 1) till the end of follow-up period (4 weeks after the last administration of the drug (day 50)
Arm/Group | BCD-066 1 µg/kg | Aranesp 1 µg/kg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 5/28 | 16/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-066 1 µg/kg (N=28) | Aranesp 1 µg/kg (N=28)
monocytes count increase (Blood and lymphatic system disorders) | 2 | 1
thrombocytes count increase (Blood and lymphatic system disorders) | 2 | 5
Hematocrit decrease (Blood and lymphatic system disorders) | 0 | 3
Hemoglobin decrease (Blood and lymphatic system disorders) | 0 | 1
WBC decrease (Blood and lymphatic system disorders) | 0 | 2
Neutrophis count decrease (Blood and lymphatic system disorders) | 1 | 3
RBC decrease (Blood and lymphatic system disorders) | 0 | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03693950/SAP_001.pdf
  • Study Protocol (2016-10-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03693950/Prot_003.pdf